CLINICAL TRIAL: NCT06636890
Title: Correlation Analysis of Xpert Carba-R Detection of Non-Colonized Carbapenem-Resistant Enterobacteriaceae in Bronchoalveolar Lavage and Rectal Swabs From Patients With Lower Respiratory Tract Infections
Brief Title: Correlation Analysis of Xpert Carba-R Detection of Non-colonized CRE in BALF and Rectal Swabs From Patients With LRTI
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-697
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae; Lower Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — The investigators will perform bronchoscopy and collect bronchoalveolar lavage fluid (BALF) samples at the time of patient enrollment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess the correlation between Xpert Carba-R detection of carbapenemase gene types in bronchoalveolar lavage samples and rectal swab samples from non-colonized CRKP patients with lower respiratory tract infections, and evaluate the relationship between first-time lower respiratory tract infections and intestinal colonization of CRKP.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* CRKP is cultured from lower respiratory tract specimens in 15 days
* Lower respiratory tract infection based on at least two of the followings: abnormal temperature (body temperature greater than 38.5°C or less than 36.5°C), leucocyte count abnormality (leucocyte count greater than 10*10^9/L or less than 4*10^9/L), and the presence of purulent tracheal secretions.

Exclusion Criteria:

* There are other bacteria that can produce carbapenemases exist in lower respiratory tract specimens
* Infected with CRE before

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population description specifies individuals diagnosed with LRTI (Lower Respiratory Tract Infection) who were enrolled based on culture-confirmed CRKP（Carbapenem-resistant Klebsiella pneumoniae）.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The detection of the carbapenemase gene types produced by Klebsiella pneumoniae in rectal swabs and BALF by Xpert Carba-R | Up to 2 weeks after each enrollment
  The investigators use the Xpert Carba-R to detect the carbapenemase gene types produced by Klebsiella pneumoniae in rectal swabs and bronchoalveolar lavage fluid (BALF) . The investigators will compare the consistency of results between the two specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- he First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China